CLINICAL TRIAL: NCT00051701
Title: Phase I/II Study of CAMPATH in Patients With Relapsing or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM.NHL232; BLA 99-0786
Record Dates: First submitted 2003-01-15; First posted 2003-01-17 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Non-Hodgkins Lymphoma
Keywords: Non-Hodgkins lymphoma; NHL; Campath; alemtuzumab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Alemtuzumab

INTERVENTIONS:
Drug: alemtuzumab

SUMMARY:
The purpose of this study is to determine the optimal dose of Campath for patients with relapsing or refractory (failed standard therapy) non-Hodgkin's lymphoma. The study will also evaluate the safety of the drug and whether it is effective in treating these patients.

DETAILED DESCRIPTION:
This study is being conducted in 2 parts with the primary objective of part 1 being to determine the maximum tolerated dose (MTD) of CAMPATH (alemtuzumab, MABCAMPATH, CAMPATH) administered intravenously (IV) once a week as treatment for relapsing or refractory non-Hodgkin's lymphoma (NHL). The primary objective of part 2 is to determine the overall response rate (complete response, CR/unconfirmed , plus partial response) of weekly IV CAMPATH in the treatment of relapsing or refractory NHL. This is a Phase I/II study, open-label, multicenter study to evaluate the efficacy and safety of weekly IV CAMPATH as therapy for patients with relapsing or refractory non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria: Patients must have:

* Pathologically confirmed diagnosis of relapsing or refractory non-Hodgkin's lymphoma that has failed conventional therapy.
* Measurable disease (lesions that can be accurately measured by CT scan and a greatest transverse diameter larger or equal to 1 cm or palpable lesions that both diameters larger or equal to 2 cm).
* Life expectancy of at least 12 weeks. - World Health Organization (WHO) performance status (PS) of 0, 1, or 2.
* Adequate marrow and organ function (details are listed in the protocol).
* Female patients with childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment. Male and female patients must agree to use an effective contraceptive method while on study treatment, if appropriate, and for a minimum of 6 months following study therapy.
* Signed, written informed consent.

Exclusion Criteria: Patients must not have:

* Prior autologous bone marrow or stem cell transplant within 6 months of study entry.
* A history of prior allogeneic bone marrow transplant or organ transplant.
* Previously untreated non-Hodgkin's lymphoma.
* Previously treated with CAMPATH.
* Patients with bulky disease, ie any single mass > 7.5cm.
* Prior radiotherapy to the only site of measurable disease.
* Medical condition requiring chronic use of oral, high-dose corticosteroids.
* Autoimmune thrombocytopenia.
* Use of investigational agents within previous 30 days or any anti-cancer therapy within the previous 3 weeks. Patients must have recovered from all acute toxicities of any prior therapy.
* Past history of anaphylaxis following exposure to humanized monoclonal antibodies.
* Active, uncontrolled infection, including human immunodeficiency virus (HIV) positive.
* Active secondary malignancy.
* Active central nervous system (CNS) involvement with NHL.
* Pregnant or lactating women. Male or female patients who do not agree to use effective contraceptive method(s) during the study.
* Any significant concurrent disease or illness that would, in the opinion of the investigator, compromise patient safety or compliance, or interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61
Dates: Start 2002-12; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (17):
- United States (17):
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Santa Fe, New Mexico
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Dallas, Texas
  - Fort Worth, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Spokane, Washington
  - Vancouver, Washington